CLINICAL TRIAL: NCT06053125
Title: The Role of Adipose Tissue in Adaptive Responses to Exercise
Brief Title: A Study of Adipose Tissue in Adaptive Responses to Exercise
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hawley E. Kunz, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-002049; K01DK134765 (NIH)
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Obesity
Keywords: exercise; adipose; cytokines
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Older adults with obesity (Experimental): Participants with obesity as determined by the principal investigator and aged 65-85 years will have an adipose tissue biopsy taken from the abdomen before and after exercise.
  Interventions: Procedure: Adipose Tissue Biopsy; Behavioral: Exercise
- Older adults without obesity (Experimental): Participants with obesity as determined by the principal investigator and aged 65-85 years will have an adipose tissue biopsy taken from the abdomen before and after exercise.
  Interventions: Procedure: Adipose Tissue Biopsy; Behavioral: Exercise
- Young adults with obesity (Experimental): Participants with obesity as determined by the principal investigator and aged 18-35 years will have an adipose tissue biopsy taken from the abdomen before and after exercise.
  Interventions: Procedure: Adipose Tissue Biopsy; Behavioral: Exercise
- Young adults without obesity (Experimental): Participants with obesity as determined by the principal investigator and aged 18-35 years will have an adipose tissue biopsy taken from the abdomen before and after exercise.
  Interventions: Procedure: Adipose Tissue Biopsy; Behavioral: Exercise

INTERVENTIONS:
Procedure: Adipose Tissue Biopsy — Fat sample collected from abdomen before exercise, immediately after exercise, and 3 hours after exercise
Behavioral: Exercise — 30 minutes of exercise on a cycle ergometer exercise machine

SUMMARY:
The purpose of this research is to determine how exercise affects fat (adipose) tissue and how changes to adipose tissue that occur during and after exercise might improve health in aging and obesity.

DETAILED DESCRIPTION:
Adipose tissue has important endocrine functions that influence metabolic health. Early evidence shows that adipose adapts to physiological stress, including exercise. The objective here is to determine how exercise-induced alterations in adipose tissue cellular composition and endocrine signaling may contribute to the beneficial adaptations to exercise in aging and obesity.

Immune cell populations and inflammatory signatures will be assessed in subcutaneous abdominal adipose tissue biopsies collected from obese and normal weight young and older adults before, immediately after, and 3 hours after a 30-min bout of cycling exercise at 70% of maximal oxygen consumption (VO2max). Mass spectrometry, Olink targeted inflammation assays, and RNA sequencing will be used for full proteomic and transcriptomic characterization of the adipose tissue secretome (the proteins and molecules secreted from the adipose tissue) and the cargo of extracellular vesicles isolated from plasma and media collected from cultured human adipose tissue explants generated from each time point.

Overall, the primary hypothesis of the proposed work is that a single bout of exercise triggers transient changes in adipose tissue paracrine/endocrine signals and immune cellular composition. The investigators propose that these responses contribute to the beneficial effects of exercise locally and in distal tissues and that the cumulative effects of acute changes in adipose tissue likely contribute to the positive alterations in adipose tissue associated with exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-35 OR 65-85.
* BMI 18.5 kg/m2 - 40 kg/m2
* Weight stable (≥ 3 months)
* Generally healthy

Exclusion Criteria:

* Participation in ≥ 30 minutes of structured physical activity ≥ 2 days per week.
* Smoking/tobacco use.
* Alcohol/substance abuse.
* Pregnancy and breastfeeding.
* Anemia.
* Abnormal renal function.
* Blood clotting disorders.
* Coronary artery disease.
* Uncontrolled thyroid disease.
* Liver disease.
* Use of medications known to influence the main outcomes of the study.
* Orthopedic problems that may be aggravated by exercise.
* Chronic disease at the discretion of the investigators.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adipose lymphocyte populations | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  The numbers of lymphocytes in the adipose tissue will be assessed by flow cytometry.
IL6 secreted from adipose tissue measured using the Olink Target Inflammation Panel (includes 96 inflammation-associated proteins) | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  The concentration of 96 IL6 will be measured using the targeted inflammation Olink proximity extension assay panel in media obtained from cultured adipose tissue explants. Adipose tissue samples will be cultured for 3 hours, and the culture media will be removed for the assessment of secreted inflammatory proteins. T
Adipose tissue macrophage populations | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Numbers of macrophages in the adipose tissue will be assessed by immunohistochemistry.
Adipose tissue gene expression of interleukin (IL)-6 measured by polymerase chain reaction (PCR). | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the inflammatory cytokine IL-6 will be measured in adipose tissue samples using real time (RT)-PCR.
Adipose tissue gene expression of interleukin (IL)-8 measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the inflammatory cytokine IL-8 will be assessed in adipose tissue samples using real-time (RT)-PCR.
Adipose tissue gene expression of cluster of differentiation 68 (CD68) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the macrophage marker CD68 be assessed in adipose tissue samples using real time (RT)-PCR.
Adipose tissue gene expression of cluster of differentiation 163 (CD163) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the anti-inflammatory macrophage marker CD163 will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of cluster of differentiation 206 (CD206) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the anti-inflammatory macrophage marker CD206 will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of adhesion G-protein coupled receptor E (ADGRE) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the macrophage marker ADGRE will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of inducible nitric oxide synthase (INOS) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the pro-inflammatory macrophage marker INOS will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of monocyte chemoattractant protein-1 (MCP1) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the inflammatory cytokine MCP1 will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of tumor necrosis factor alpha (TNFa) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the inflammatory cytokine TNFa will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of leptin (LEPD) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the pro-inflammatory adipokine LEPD will be assessed in adipose tissue samples using RT-PCR.
Adipose tissue gene expression of adiponectin (ADIPOQ) measured by PCR. | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Gene expression of the anti-inflammatory adipokine ADIPOQ will be assessed in adipose tissue samples using RT-PCR.
Inflammatory proteins found in adipose tissue measured using the Olink Target Inflammation Panel (includes 96 inflammation-associated proteins) | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  The concentrations of 96 different inflammatory proteins (including various cytokines and adipokines) will be measured in adipose tissue lysates using the targeted inflammation Olink proximity extension assay panel. This assay measures all 96 proteins in a single assay and all are reported as normalized protein expression values.
Protein cargo of adipose extracellular vesicles measured using mass spectrometry | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Adipose tissue samples will be cultured for 3 hours, and the culture media will be removed. From this media, extracellular vesicles will be isolated. In these extracellular vesicles, mass spectrometry will be performed to examine the entire proteome (all proteins) contained within these extracellular vesicles. Using the large number of proteins identified, the investigators will examine changes in categories of protein types (e.g., inflammatory proteins, metabolic proteins, transcriptional proteins).

SECONDARY OUTCOMES:
Adipocyte cell size | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Adipocyte cell size will be determined using methylene blue staining and microscopy.
Plasma IL6 concentrations measured using the Olink Target Inflammation Panel | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  The concentration of IL6 will be measured in plasma samples using the targeted inflammation Olink proximity extension assay panel. This assay measures 96 proteins in a single assay and all are reported as normalized protein expression values.
Protein cargo of plasma extracellular vesicles measured using mass spectrometry extracellular vesicles | Pre-exercise, immediately post-exercise, and 3 hours after exercise
  Extracellular vesicles will be isolated from plasma samples. In these extracellular vesicles, mass spectrometry will be performed to examine the entire proteome (all proteins) contained within these extracellular vesicles. Using the large number of proteins identified, the investigators will examine changes in categories of protein types (e.g., inflammatory proteins, metabolic proteins, transcriptional proteins).

OTHER OUTCOMES:
Body fat percentage | Baseline
  Body fat percentage will be assessed using dual energy x-ray absorptiometry (DEXA).
Cardiorespiratory Fitness | Baseline
  Individual maximal oxygen consumption (VO2 max) will be assessed by indirect calorimetry during a graded exercise test
White blood count | Baseline
  White blood count with differential will be measured by the Mayo clinical lab.
Fasting plasma insulin | Baseline
  Plasma insulin will be measured by the Mayo Clinical Lab.
Fasting plasma glucose | Baseline
  Plasma glucose will be measured by the Mayo Clinical Lab.
Hemoglobin A1c (HbA1c) | Baseline
  HbA1c will be measured by the Mayo Clinical Lab.

CONTACTS AND LOCATIONS:
Overall Officials: Hawley Kunz, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials